CLINICAL TRIAL: NCT05898789
Title: Pragmatic Hybrid Type 1 Effectiveness-implementation (E-I) Trial of a Virtual Cancer Rehabilitation Program
Brief Title: Virtual Rehabilitation for Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-6035
Record Dates: First submitted 2023-05-07; First posted 2023-06-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer, Stage 0; Colorectal Cancer Stage I; Head and Neck Cancer Stage I; Lymphoma; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Colorectal Cancer Stage II; Colorectal Cancer Stage III; Head and Neck Cancer Stage II; Head and Neck Cancer Stage III; Lymphoproliferative Disorders
MeSH Terms: conditions — Breast Carcinoma In Situ; Colorectal Neoplasms; Head and Neck Neoplasms; Lymphoma; Breast Neoplasms; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaRE@Home intervention (Experimental)
  Interventions: Behavioral: CaRE@Home intervention
- Usual Care group (No Intervention)

INTERVENTIONS:
Behavioral: CaRE@Home intervention — participants randomized to the intervention arm will complete a virtual 8 week exercise and education program.
  Arms: CaRE@Home intervention

SUMMARY:
Pragmatic hybrid type 1 effectiveness-implementation (E-I) trial of a virtual cancer rehabilitation program: The study team will conduct a multi-center hybrid type I effectiveness-implementation study to examine the clinical effectiveness and implementation potential of an 8-week multidimensional virtual cancer rehabilitation intervention (CaRE@Home) for cancer survivors with identified cancer-related impairments on level of overall disability (primary outcome) and patient reported physical and social functioning, anxiety, work status, quality of life, and physiologic changes (secondary outcomes). The study team will conduct a multi-centre pragmatic randomized controlled trial (RCT) (Vancouver, Toronto, Saint John and St. John's) to evaluate effectiveness and using the CIFR, the study team will identify potential factors that may affect successful implementation and integration of CaRE@Home in different cancer settings.

DETAILED DESCRIPTION:
Comprehensive multidimensional rehabilitation programs that include both exercise and self management education have the potential to concurrently improve a wide range of post treatment side-effects and overall patient function. In 2017, the Cancer Rehabilitation and Canadian Cancer Rehabilitation (CanRehab) Team: Improving the systematic identification, management, and treatment of the adverse effects of cancer.

Survivorship program at Princess Margaret Cancer Centre launched an evidence driven group based multidimensional Cancer Rehabilitation and Exercise program (CaRE@ELLICSR) for patients who have identified cancer-related impairments. The 8-week program integrates a number of evidence-based techniques to sustain behavioural change and consists of weekly1-hr group exercise classes followed by 1-hr self-management skills education delivered by a rehabilitation expert. Participants return for follow-up at 3 and 6 months post-intervention to monitor progress and adapt exercise as needed. CaRE@ELLICSR has resulted in improvements in overall levels of disability, social functioning, distress, and physical activity. Program satisfaction is high, and wait times are within the target of <1 month. However, access is an issue with ~50% of referred patients unable to participate due to travel distance, transportation costs or competing obligations (unpublished data).

To increase access, a virtual on-line version of the CaRE program (CaRE@Home) was developed using a series of iterative steps proposed by the NCI Research-Tested Intervention Programs.

The CaRE@Home program is currently undergoing single-group feasibility pilot testing (completion Oct 2019, funded by Ontario Institute for Cancer Research). Feasibility outcomes collected to date demonstrate high program acceptability with 95% of referred patients enrolled and 94% program adherence. The final steps of this process are to formally evaluate effectiveness and prepare for real-world implementation, which is the focus of Project Two of this application. If effective, the virtual CaRE@Home program has the potential to extend access to critical cancer rehabilitation services to a greater number of cancer survivors in need. It also has immense potential to be adapted and scaled to other centres that lack the resources required to deliver in-house cancer rehabilitation services. In Project Two the study team will conduct a multi-center hybrid type I effectiveness-implementation study to examine the clinical effectiveness and implementation potential of CaRE@Home for cancer survivors with identified cancer-related impairments.

Principal Research Aims:

Aim 2.1: Test the effectiveness of CaRE@Home vs. usual care (UC) on disability (primary outcome) and patient reported and physiological outcomes (secondary outcomes) at 3-months post-intervention.

Aim 2.2: Conduct a descriptive implementation-focused process evaluation to inform future implementation efforts

Methods The project is a hybrid type 1 effectiveness-implementation (E-I) study. The aim of hybrid trials are to better align research and practice and to provide a pathway for rapidly moving knowledge from research to implementation. In hybrid type 1 studies, the primary aim is to determine effectiveness in the setting where it will be implemented and the secondary aim is to better understand the context for implementation. This methodology promotes the study of implementation as early as possible in the research process and can serve a dual purpose in helping to explain effectiveness results and informing future implementation efforts.

Aim 2.1: Effectiveness evaluation of CaRE@Home (months 36-58) Design: The study team will conduct a multi-centre pragmatic RCT (Vancouver, Toronto, Saint John and St. John's) to evaluate effectiveness. Clinical effectiveness studies place a greater emphasis on external validity and generalizability than efficacy trials and typically include heterogeneous patient populations and settings. Participants will be randomized into CaRE@Home or UC.

Recruitment and Data Collection: Eligible participants will be identified by their oncology team, and provided information about the study along with contact information for the local study team. Depending on timing, the ePSM platform (Project One) may also be used to identify and invite potential participants. Interested patients will be pre-screened by telephone (eligibility tools above), and those who are eligible will be invited to an in-person baseline assessment (T1). Site-specific screening logs will be maintained. At the baseline assessment, participants will provide consent and complete PRO and physiological measures (see below) with a trained assessor. Following the assessment, the research assistant will obtain the randomization assignment. Those assigned to CaRE@Home will be registered into the CaRE@Home platform.

Follow-up assessment for both groups will occur at 8-weeks (T2 immediate post intervention) and 3 months post-intervention (T3). The CaRE@Home group will have an additional 6 months post-intervention (T4) to assess maintenance. Randomization: Permuted block randomization, with stratification by center and on/finished treatment will allocate participants to either CaRE@Home or UC. Randomization will be computer-generated and managed by the Department of Biostatistics at Princess Margaret Cancer Centre.

Description of Study Arms: i) Care@Home is an 8-week program comprised of: 1) weekly e-modules providing interactive education to promote self-management skills; 2) individualized progressive exercise prescription supported with mobile application (PhysitrackTM); 3) wearable technology (FitbitTM) to track activity and sleep; and 4) weekly brief telephone counselling with a member of the rehabilitation team (see Appendix 4 CaRE@Home program elements). Informed by behavior change theory, the program elements aim to provide patients with the knowledge and tools needed to reach and maintain their wellness and exercise goals. Training for health professionals: In person assessments and weekly phone calls will be delivered by a rehabilitation/exercise professional who has experience working with cancer survivors. The exercise professionals will receive comprehensive training and ongoing supervision. Training will be provided by a Motivational Interviewing Network of Trainers certified trainer (Dr. M. Obadia). The training will be videotaped and an online tool box with training resources will be developed to support future scalability. ii) UC will receive usual care and will be asked to complete in-person assessment at T2 and T3. Following T3 assessment, the UC group will be offered the CaRE@Home program.

Data analysis: Demographic and clinical information across all time points will be summarised using descriptive statistics and plotted across all time points. Effectiveness will be assessed on the full set of consented participants in accordance with the intention to treat principle. The primary outcome is the difference in WHODAS 2.0 mean score between CaRE@Home and UC at T3. Differences on secondary outcomes at T3 will also be compared between the two treatment arms using paired t test or paired Wilcoxon rank-sum test. Maintenance of treatment gains in the CaRE@Home group will be analyzed at T4. An estimate of the effect size and parameters and corresponding confidence intervals will be calculated between groups at T3 and over time (within groups). Variability of the main and interaction effects will be examined on the primary clinical outcome (WHODAS 2.0) and each of the secondary outcomes using separate longitudinal analysis models such as mixed model regression and generalized estimating equation models. Sensitivity analysis will be conducted, adjusting for important clinical factors using the regression model. Finally, a cost-utility analysis will be undertaken to estimate the incremental cost per quality-adjusted life year (QALY) of the intervention arm compared to the control arm.

Sample Size: Our sample size calculations is based on 80% power with a two-sided alpha-level at 0.05 and an estimated effect size of 0.4 standard deviation of the primary endpoint.

Assuming attrition of up to 30% and adherence to be 80%, 388 patients will be recruited (or 194 patients per arm). The number of potentially eligible patients across sites is estimated to be 170 patients per month. Based on proposed staffing per site, a maximum of 20 patients can be enrolled per month in Toronto/Vancouver and 10 per site in NB/NFLD. Enrollment is estimated to take 6-7 months. The study team will use multiple strategies to promote retention and prevent attrition.

Aim 2.2: Implementation-focused Process Evaluation (months 30-52) Design: In order to inform the implementation of CaRE@Home, a process evaluation will be conducted and guided by the RE-AIM framework[88]. The CFIR will be used to examine context and understand relevant barriers and facilitators across and within CanRehab sites. See Table 3 for Implementation Framework/Process Evaluation Questions and Tools.

Data Collection Tools: Data tools will include interviews/focus groups, surveys, screening logs, observational notes, technical reports, infrastructure review to inform costs as well as staffing and infrastructure requirements. The study team will triangulate the data from the different quantitative and qualitative sources to answer questions developed based on elements of the selected frameworks and summarize our findings.

Data Analysis: Descriptive variables will be presented as means, distributions, and proportions with differences between subgroups compared. Qualitative information from open-ended survey questions, interviews, and research log entries will be transcribed and analyzed using common deductive qualitative analysis techniques[133] following the CFIR qualitative data analysis templates. Following this, all transcripts will be coded and additional inductive codes will be added.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18 years or older
* 2) Diagnosed with breast (stage 0-III), colorectal (stage I-III), head and neck (stage I-III), or lymphoma/lymphoproliferative disorder (excluded: recurrent, refractory, progressive, received or planning to receive transplant)
* 3) Completed a primary treatment (i.e. surgery and/or radiation and/or systemic therapy of any kind) within the last 24 months
* 4) If patients received systemic therapy of a fixed duration with adjuvant/curative intent, the main part should be completed, but patients are eligible if on primary, maintenance, or other adjuvant systemic therapy (e.g. eligible while on trastuzumab, immunotherapy, rituximab, oral endocrine or targeted therapy - ie ibrutinib). Indolent non-curative lymphoma patients are eligible if they have response to systemic therapy
* 5) Communicate sufficiently in English to complete intervention and questionnaires
* 6) Willing to be randomized and participate in the intervention and in-person assessments; 6) Internet access
* 7) An indication for cancer rehabilitation (WHO-DAS score >5).

Exclusion Criteria:

* 1) Impaired functional status that would preclude rehabilitation (PRFS >3)
* 2) Indication of major depressive disorder (PHQ-2 >3)
* 3) Diagnosis of neurological disease or condition significantly limiting cognitive functioning, such as language or memory (e.g., Alzheimer's disease or other dementia, severe traumatic brain injury);
* 4) Conditions or current injuries which are not appropriate for distance based exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Disability | 6 months
  measured using the World Health Organization Disability Assessment Schedule 2.0, which is a cross-cultural standardized method for measuring limitations and restrictions on individuals' activities and participation in society. The average scores are comparable to the WHODAS 5-point scale, he total score for WHODAS ranges from 0-100, where a high score indicates major living limitations ((0-0.49) = none, mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4).

SECONDARY OUTCOMES:
Demographics | 6 months
  Demographic details will be collected from participants at the time of initial assessment via an intake questionnaire. There are no scales, only patient reported outcome questions
Physical functioning | 8 months
  Measured using the 10-item sub-scale of the short form Health Survey (scale from 0 (negative health) to 100 (positive health))
Social functioning | 8 months
  Measured using the Social Difficulties Inventory. A zero score indicates perfect comparison with consensus group and > or equal to 2 indicates unacceptable performance/remedial action required.
Anxiety | 8 months
  Measured using the Generalized Anxiety Disorder 7. The overall GAD 7 score ranges between 0-21, with zero meaning no anxiety and 21 meaning severe anxiety.
Physical activity | 8 months
  Measured using the the International Physical Activity Questionnaire - Short Form. It assesses the number of days/time spent on PA in moderate intensity, vigorous intensity, walking of at least 10-min duration the last 7 days, and time spent sitting on weekdays the last 7 days.
Work functioning | 8 months
  measured using the short version of the World Health Organization's Heath and Work Performance Questionnaire. Absenteeism is scored in terms of hours lost per month, which is to say that a high score indicates a higher amount of absenteeism. The measure of absolute absenteeism is expressed in raw hours, with a negative lower bound (if the person works more than expected) and an upper bound equal to the number of hours the respondent is expected to work. The measure of relative absenteeism is expressed as a percentage of expected hours and ranges between a negative number (works more than expected) and 1.0 (always absent).
Health status | 8 months
  measured using the EuroQol 5D-5L[81], a brief and frequently used measure of health status that consists of a weighted sum of five dimensions: Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression, and provides a simple descriptive profile and a single index value for health status.
Safety status | 8 months
  assessed throughout the study and any adverse events resulting from the intervention will be scored on the CTCAE version 5.0[82] and documented during the health coaching calls and physical assessments with the exercise professional.
Physiological measure of height | 8 months
  Participant height at baseline
Physiological measure of weight | 8 months
  Participant weight at all physical assessments (T1, T2, T3, T4) will be collected. The data will inform calculations for BMI.
Physiological measures of cardiorespiratory fitness | 8 months
  Measured with the six minute walk test (6MWT)
Grip strength | 8 months
  Physiological measure of muscular strength measured with hand grip strength and measured bilaterally with standard Jamar dynamometer.Per CSEP protocol, an average of 2 trials with a 2 min rest in-between trials will be taken. The best of the left and right hand will be taken as the overall grip score. Participant handedness will also be recorded.
30-second sit to stand test | 8 months
  Physiological measure of endurance is measured with the 30-second sit to stand test for lower body strength
Physiological measures of performance | 8 months
  Measured with the 4-meter Gait speed test

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, PhD, Principal Investigator — UHN Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada